CLINICAL TRIAL: NCT06211153
Title: Real-world Effectiveness of Asciminib and Treatment Patterns in Patients With Chronic Myeloid Leukemia With T315I Mutation - a Chart Review Study of Patients Treated in the Asciminib Managed Access Program (MAP)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A2004
Record Dates: First submitted 2023-12-15; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Chronic Myeloid Leukemia With T315I Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Asciminib

SUMMARY:
This non-interventional study (NIS) was a retrospective chart review analyzing existing data from patients participating in the asciminib MAP.

ELIGIBILITY:
Study Population: Key Inclusion/Exclusion Criteria Inclusion criteria

* Diagnosis of CML (chronic phase, accelerated phase or blast crisis).
* Confirmed presence of T315I mutation prior to asciminib initiation.
* Patients enrolled in the asciminib MAP and received their first dose of asciminib between 01 November 2018 and 30 April 2022. Patients must have received at least one dose of asciminib.
* Appropriate approval was obtained for the patient chart review including:

  * Patient signed the informed consent form (ICF) or,
  * Individual ICF waiver was granted by an institutional review board/ Independent Ethics Committee (IRB)/ IEC.

Exclusion criteria

• Age less than 18 years old at the time of initiating asciminib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Major molecular response (MMR) at 6 months | At 6 months
Major molecular response (MMR) by 6 months | By 6 months

SECONDARY OUTCOMES:
MMR at and by 3, 9, and 12 months | At and by 3, 9, and 12 months
Complete cytogenic response (CCyR) at and by 3, 6, 9, and 12 months | At and by 3, 6, 9, and 12 months
Complete hematologic response (CHR) at and by 3, 6, 9, and 12 months | At and by 3, 6, 9, and 12 months
Time to first CCyR at and by 3, 6, 9, and 12 months | At and by 3, 6, 9, and 12 months
Gender | Baseline
Race | Baseline
Time from CML diagnosis to study index (i.e., asciminib) start date | Baseline
Country of residence | Baseline
Status of CML at baseline | Baseline
Number of patients per response type at asciminib start date | Baseline
  Response types were MMR, CCyR, and CHR.
Stem-cell transplant performed status | Baseline
Medical history by system-organ-class, preferred term from CML diagnosis to asciminib start date | Baseline
Overall tyrosine kinase inhibitors (TKIs) prior to index date | Baseline
Prior TKIs between CML diagnosis and T315I mutation diagnosis | Baseline
Prior TKIs between T315I mutation diagnosis and index date | Baseline
Sequence of prior TKI treatment patterns | Baseline
Number of patients with response to prior TKIs from CML diagnosis to asciminib (index date) | Baseline
  Response types were MMR, CCyR, and CHR.
Number of patients with response to prior TKIs between CML diagnosis to T315I mutation diagnosis | Baseline
  Response types were MMR, CCyR, and CHR.
Number of patients with response to prior TKIs between T315I mutation diagnosis to asciminib start (index date) | Baseline
  Response types were MMR, CCyR, and CHR.
Number of patients with intolerance to prior TKIs, per category | Baseline
  Categories were discontinuation due to adverse events, relationship to treatment, and outcome.
Number of patients with intolerance to last TKI prior to asciminib, per category | Baseline
  Categories were discontinuation due to adverse events, relationship to treatment, and outcome.
Asciminib dose | Up to 13 months
Asciminib discontinuation | Up to 13 months
Duration of exposure to asciminib | Up to 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Basel, Switzerland